CLINICAL TRIAL: NCT05765604
Title: A Randomized, Parallel Controlled, Double-blind, Single-center Phase I Clinical Trial of Recombinant COVID-19 Variant Vaccine (Sf9 Cell)(WSK-V102) in People Aged 18 Years or Older
Brief Title: Phase I Clinical Trial of Recombinant COVID-19 Variant Vaccine (Sf9 Cell) (WSK-V102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WSKCT001
Record Dates: First submitted 2023-03-10; First posted 2023-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): low dose and high dose, only one dose at day 0
  Interventions: Biological: Recombinant COVID-19 variant vaccine(Sf9 cell)
- control group (Active Comparator): one dose at day 0
  Interventions: Biological: Recombinant COVID-19 vaccine(CHO cell)

INTERVENTIONS:
Biological: Recombinant COVID-19 variant vaccine(Sf9 cell) — IM
  Arms: test group
Biological: Recombinant COVID-19 vaccine(CHO cell) — IM
  Arms: control group

SUMMARY:
Subjects aged 18 and above who have been completed primary or booster vaccination of COVID-19 inactivated vaccines for 3 months or more, to conduct a randomized, parallel controlled, double-blind, single-center phase I clinical trial of Recombinant variant COVID-19 vaccine (Sf9 cell)(WSK-V102) to evaluate the safety, tolerance and immunogenicity of this vaccine in the study population.

DETAILED DESCRIPTION:
Low and high doses of study vaccine were compared with control groups to evaluate the safety and immunogenicity of the study vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. Obtain the subject's informed consent and sign the informed consent form.
3. The subject is able and willing to comply with the requirements of the clinical trial protocol and is willing and able to comply with all study plan contents and other requirements of the study.
4. Armpit body temperature < 37.3℃.
5. People who have had basic or enhanced immunization with COVID-19 vaccine for 3 months or more;
6. SARS-CoV-2 nucleic acid screening was negative in the last 24 hours.
7. Anti-sars-cov-2 IgM antibody was negative during the screening period.
8. BMI of 18.5-30.0 kg/m2.
9. Women's non-pregnancy period (pregnancy test results are negative), non-lactation period.
10. Fertile Women (WOCBP) subjects had taken effective contraceptive measures 1 month before enrollment.
11. WOCBP subjects and male subjects, who do not plan to become pregnant for 6 months from the screening period to the last dose of immunization, agree to take effective contraceptive measures for 6 months from the screening visit to the last dose of immunization.
12. WOCBP subjects and male subjects agree not to donate eggs (oocytes, oocytes) for assisted reproduction (WOCBP subjects) or to refrain from sperm donation (male subjects) for a period of 6 months from screening visit to the last dose of immunization.
13. Subjects eligible for immunization with this product after medical history, physical examination and clinical judgment of health.

Exclusion Criteria:

1. Have cancer; Or have other serious chronic diseases such as uncontrolled asthma, diabetes, liver and kidney disease, thyroid disease, convulsions, epilepsy and other neurological/psychiatric disorders.
2. have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukaemia or other autoimmune disease;
3. Those who are allergic to any component of the experimental vaccine have had a history of severe vaccine allergic reaction in the past.
4. History of SARS or MERS or SARS-CoV-2 infection/illness within 3 months.
5. Patients with more serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension that cannot be controlled by drugs.
6. Congenital or acquired angioedema/neuroedema.
7. Urticaria in the year prior to receiving the experimental vaccine.
8. asplenia or functional asplenia.
9. Thrombocytopenia or other clotting disorders (which may cause intramuscular injection contraindications).
10. Needle fainter.
11. Immunosuppressive therapy, antiallergy therapy, cytotoxic therapy, and inhaled corticosteroids (excluding corticosteroid spray for allergic rhinitis and topical corticosteroids for acute non-concurrent dermatitis) for 14 or more days within 6 months prior to receiving the experimental vaccine.
12. Received blood products within 3 months prior to receiving the trial vaccine.
13. Received other investigational drugs within 1 month prior to receiving the experimental vaccine.
14. Received subunit or inactivated vaccine within 14 days or live attenuated vaccine within 1 month prior to receiving the experimental vaccine.
15. are receiving anti-TB treatment.
16. Medical, psychological, social or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's signing of informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
solicited adverse events (AE) | 0-14 days after vaccination
  Incidence of solicited adverse events (AE)

SECONDARY OUTCOMES:
laboratory safety | 3 days after vaccination
  Changes in laboratory tests on day 3 after vaccination
safety outcome | 30 days after vaccination,12 months after vaccination
  Incidence of unsolicited adverse events (AE) and serious adverse events (SAE)
binding antibodies | 14 days, 30 days, 3 months and 6 months
  Geometric mean Titer (GMT) and Geometric mean growth multiple (GMFI) of S-RBD protein-specific antibodies (ELISA) against SARS-CoV-2
neutralizing antibodies | 14 days, 30 days, 3 months and 6 months
  Geometric mean Titer (GMT) and Geometric mean growth multiple (GMFI) of neutralizing antibodies against SARS-CoV-2 prototype strain and Omicron variant strain (according to the prevailing strain)
cellular immune | 14 days and 3 months
  ELISpot was used to detect the cell frequencies of IFN-γ and IL-2 secreted by SARS-CoV-2 S-RBD protein

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease Control, Taizhou, China